CLINICAL TRIAL: NCT03861806
Title: Reliability of Paired Associative Stimulation-induced Neuroplasticity After Stroke
Acronym: PASS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Burke Medical Research Institute (Other)
Responsible Party: Principal Investigator, Tomoko Kitago, Lab Director, Burke Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HMRL-001
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: We plan a randomized crossover study of sham and true PAS.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAS true (Experimental): Participants will receive paired associative stimulation therapy with a modulatory inter-stimulus interval.
  Interventions: Behavioral: PAS true
- PAS sham (Sham Comparator): Participants will receive paired associative stimulation therapy with a non modulatory inter-stimulus interval.
  Interventions: Behavioral: PAS sham

INTERVENTIONS:
Behavioral: PAS true — Participants will receive paired associative stimulation (transcranial magnetic stimulation and peripheral nerve stimulation) with an inter-stimulus interval length known to modulate corticospinal excitability.
  Arms: PAS true
Behavioral: PAS sham — Participants will receive paired associative stimulation (transcranial magnetic stimulation and peripheral nerve stimulation) with an inter-stimulus interval length known to not modulate corticospinal excitability.
  Arms: PAS sham

SUMMARY:
Paired associative stimulation (PAS) is a non-invasive stimulation method which is known to modulate corticospinal excitability through mechanisms related to long-term potentiation and long-term depression. The purpose of this study is to determine the reliability of individual subject's response (i.e., change in corticospinal excitability) to PAS in patients with chronic stroke (>6 months) with upper limb motor deficits.

DETAILED DESCRIPTION:
One of the assumptions in stroke rehabilitation is that motor training will lead to motor re-learning and persistent improvements through mechanisms involving neuroplasticity, defined as the ability of the brain to change its structure and function in response to injury, activity, or change in environment. A way to measure a patient's capacity for neuroplasticity may be useful in guiding selection of patients for rehabilitative interventions, or to assess the effect of pharmacological agents on neuroplasticity which may aid in augmenting motor recovery. One method to assess neuroplasticity non-invasively in humans through the use of paired associative stimulation (PAS). PAS is a form of non-invasive stimulation that modulates corticospinal excitability through mechanisms related to long-term potentiation (LTP) and long-term depression (LTD). In PAS, repetitive pairing of peripheral nerve stimulation with a transcranial magnetic stimulation (TMS) pulse over the contralateral motor cortex will increase or decrease corticospinal excitability, depending on the timing between the two stimuli. In healthy subjects and patients with stroke, PAS has successfully been used to facilitate corticospinal excitability as a means to enhance motor performance. In this study, we plan to use PAS as an assay of corticospinal plasticity rather than as a therapeutic intervention in patients with chronic motor deficits (>6 months) due to ischemic stroke.

There is large interindividual variability in individuals' responses to PAS, which may be useful in examining its relationship to motor learning, but the reliability of the measure will need to be assessed prior to using this measure to make inferences about a subject's general capacity to learn motor tasks. The reliability of the response to PAS and its relationship to clinical factors such as stroke severity, has not been well studied in patients with stroke. Results from a preliminary experiment suggest that stroke patients who have a robust response to facilitatory PAS on their unaffected hemisphere have more severe motor deficits than those who do not have a significant response to PAS.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ischemic stroke with residual arm weakness (Fugl-Meyer Upper Limb < 60) more than 6 months prior to enrollment.
* Ability to give informed consent and understand the tasks involved.
* Age over 18 years.

Exclusion Criteria:

* Hemorrhagic Stroke
* Contraindications to TMS: history of seizure/epilepsy, pacemaker, other neurological disorders, brain surgery, metal implant/fragment in the head, pregnancy
* Taking medications or substances that are known to affect PAS-induced plasticity within the past 2 months: selective serotonin reuptake inhibitors, dopamine, dopamine agonists, haloperidol, lithium, acetylcholinesterase inhibitors, beta-blockers, nimodipine, levetiracetam, ethosuximide, benzodiazepines, baclofen, nicotine
* Peripheral neuropathy or history of nerve injury in the paretic upper limb.
* Social and/or personal circumstances that interfere with ability to return for all study visits.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Change in motor evoked potential amplitude | Baseline, up to 30 min Post PAS
  Assessment of corticospinal excitability

CONTACTS AND LOCATIONS:
Locations (1):
- Burke Neurological Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No